CLINICAL TRIAL: NCT04259528
Title: Endoscopic Ultrasound Findings in Esophageal Atresia Following Surgical Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael A. Manfredi, MD, Medical Director of Esophageal and Airway Treatment Center, Assistent Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00032913
Record Dates: First submitted 2020-01-16; First posted 2020-02-06 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Atresia
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with esophageal stricture following surgical repair (Experimental): Patients with esophageal atresia following surgical repair who developed an esophageal stricture
  Interventions: Device: Pediatric endoscopic ultrasound

INTERVENTIONS:
Device: Pediatric endoscopic ultrasound — endoscopic ultrasound at the esophageal stricture site to assess echo texture and esophageal layers

SUMMARY:
Children with esophageal atresia who undergo surgical repair are at risk for anastomotic stricture following surgery. Esophageal stricture can be treated with serial endoscopic dilation but may ultimately need surgical resection if the stricture proves refractory to therapy. Several risk factors have been reported for development of recalcitrant stricture, but to date, no studies have specifically examined the relationship between anastomotic thickness and echotexture at time of initial postoperative endoscopy and treatment outcomes. Other risk factors that have been implicated in the development of recalcitrant stricture include gastroesophageal reflux disease, anastomotic leak, long-gap esophageal atresia, and gestational age. Moreover, it is poorly understood how esophageal layers alter and progress with repeated therapeutic dilation. The investigator hypothesize that the initial thickness and echotexture will help determine therapeutic outcome. It will also help us understand the progression of esophageal echotexture following therapeutic dilation.

ELIGIBILITY:
Inclusion Criteria:

- Patients ages 0-21 years old at time of evaluation with a suspected diagnosis of esophageal stricture secondary to esophageal atresia (with or without Tracheoesophageal fistula) post surgical repair

Exclusion Criteria:

* Patients with pre-diagnosis of eosinophilic esophagitis
* Patients with pre-diagnosis of congenital esophageal stricture
* Patients diagnosed with esophageal stricture secondary to caustic ingestion
* Patient is diagnosed with an esophageal perforation at time of endoscopy

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Predict post surgical primary repair outcome in patients with esophageal atresia using endoscopic ultrasound | 2 years
  Patients with esophageal atresia following surgical repair will undergo an endoscopic ultrasound procedure to measure esophageal layer thickness and to describe esophageal echo-texture characteristics at the anastomotic site

CONTACTS AND LOCATIONS:
Overall Officials: michael manfredi, MD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kouchi K, Yoshida H, Matsunaga T, Ohtsuka Y, Nagatake E, Satoh Y, Terui K, Mitsunaga T, Ochiai T, Arima M, Ohnuma N. Endosonographic evaluation in two children with esophageal stenosis. J Pediatr Surg. 2002 Jun;37(6):934-6. doi: 10.1053/jpsu.2002.32921. PMID 12037771
- [Background] Amae S, Nio M, Kamiyama T, Ishii T, Yoshida S, Hayashi Y, Ohi R. Clinical characteristics and management of congenital esophageal stenosis: a report on 14 cases. J Pediatr Surg. 2003 Apr;38(4):565-70. doi: 10.1053/jpsu.2003.50123. PMID 12677567
- [Result] Tambucci R, Angelino G, De Angelis P, Torroni F, Caldaro T, Balassone V, Contini AC, Romeo E, Rea F, Faraci S, Federici di Abriola G, Dall'Oglio L. Anastomotic Strictures after Esophageal Atresia Repair: Incidence, Investigations, and Management, Including Treatment of Refractory and Recurrent Strictures. Front Pediatr. 2017 May 29;5:120. doi: 10.3389/fped.2017.00120. eCollection 2017. PMID 28611969
- [Result] Khan KM, Foker JE. Use of high-resolution endoscopic ultrasonography to examine the effect of tension on the esophagus during primary repair of long-gap esophageal atresia. Pediatr Radiol. 2007 Jan;37(1):41-5. doi: 10.1007/s00247-006-0333-9. Epub 2006 Oct 17. PMID 17043852